CLINICAL TRIAL: NCT03388437
Title: Non-invasive Neurally Adjusted Ventilatory Assist Versus Nasal Intermittent Positive Pressure Ventilation for Preterm Infants After Extubation: A Randomised Control Trial
Brief Title: Non-invasive Neurally Adjusted Ventilatory Assist Versus Nasal Intermittent Positive Pressure Ventilation for Preterm Infants After Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Fahad Armed Forces Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Raniah Aljeaid, Neonatal Fellow, King Fahad Armed Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 202
Record Dates: First submitted 2017-12-16; First posted 2018-01-03 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Prematurity; Respiratory Failure; Ventilator Lung; Newborn
Keywords: Non-invasive Neurally Adjusted Ventilatory Assist NI-NAVA; Nasal Intermittent Positive Pressure Ventilation NIPPV; post extubation
MeSH Terms: conditions — Premature Birth; Respiratory Insufficiency; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
  * A web generated a block randomisation list.
  * A block of 4, stratification based on GA, gender & antenatal steriods
  * Sequentially numbered, opaque and sealed envelopes
  * Restricted access to envelopes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NI-NAVA (Experimental): Initial setting; NAVA level of 2; PEEP of 5-6 cm H 2 O, apnea time 5-10 seconds, target Edi maximum between 10-15 and minimum < 5 for 72 hours post extubation
  Interventions: Device: NI-NAVA
- NIPPV (Active Comparator): Initial setting; PIP can be increased by 2 cm H 2 O from the pre-extubation PEEP of 5-6 cm for 72 hours post extubation
  Interventions: Device: NIPPV

INTERVENTIONS:
Device: NI-NAVA — Enrolled infants will receive Surfactant and loading dose of Caffeine citrate prior to extubation. The criteria for extubation will be as per attending decision.
  The device is used Servo-I ventilator (MAQUET). FiO 2 % is adjusted to maintain oxygen saturation between 90-94% on pulse oximetry. The flow rate is 8-10 L/min. NAVA electrodes will be inserted within nasogastric catheter & positioned at the level of diaphragm.Vital signs and ventilatory parameters are monitored hourly. Blood gases will be measured before and one hour after extubation
  Arms: NI-NAVA
Device: NIPPV — Enrolled infants will receive Surfactant and loading dose of Caffeine citrate prior to extubation. The criteria for extubation will be as per attending decision.
  The device is used Servo-I ventilator (MAQUET). FiO 2 % is adjusted to maintain oxygen saturation between 90-94% on pulse oximetry. The flow rate is 8-10 L/min. NAVA electrodes will be inserted within nasogastric catheter & positioned at the level of diaphragm.Vital signs and ventilatory parameters are monitored hourly. Blood gases will be measured before and one hour after extubation
  Arms: NIPPV

SUMMARY:
Non-invasive respiratory support has been emerging in the management of respiratory distress syndrome (RDS) in preterm infants to minimise the risk of lung injury. Intermittent positive pressure ventilation (NIPPV) provides a method of augmenting continuous positive airway pressure (CPAP) by delivering ventilator breaths via nasal prongs.It may increase tidal volume, improve gas exchange and reduce work of breathing. However, NIPPV may associate with patient-ventilator asynchrony that can cause poor tolerance and risk of intubation. It may also in increased risk of pneumothorax and bowel perforation because of increase in intrathoracic pressure.

On the other hand, neurally adjusted ventilatory assist (NAVA) is a newer mode of ventilation, which has the potential to overcome these challenges. It uses the electrical activity of the diaphragm (EAdi) as a signal to synchronise the mechanical ventilatory breaths and deliver an inspiratory pressure based on this electrical activity. Comparing NI-NAVA and NIPPV in preterm infants, has shown that NI-NAVA improved the synchronization between patient and ventilator and decreased diaphragm work of breathing .

There is lack of data on the use of NI-NAVA in neonates post extubation in the literature. To date, no study has focused on short-term impacts. Therefore, it is important to evaluate the need of additional ventilatory support post extubation of NI-NAVA and NIPPV and also the risk of developing adverse outcomes.

Aim:

The aim is to compare NI-NAVA & NIPPV in terms of extubation failure in infants< 32 weeks gestation.

Hypothesis:

Investigators hypothesized that infants born prematurely < 32 weeks gestation who extubated to NI-NAVA have a lower risk of extubation failure and need of additional ventilatory support.

DETAILED DESCRIPTION:
Study Design: Randomised controlled trial

Study Setting: single center NICU level III, KFAFH tertiary care center , Jeddah Saudi Arabia

ELIGIBILITY:
Inclusion Criteria:

1. Born less than 32 weeks gestation with respiratory distress syndrome (RDS) and requiring endotracheal tube and mechanical ventilation.
2. Less than two weeks old
3. First extubation attempt
4. CRIB score 0-5
5. Written-informed parental consent for the study

Exclusion Criteria:

1. Major congenital malformations or respiratory abnormalities
2. Neuromuscular disease
3. phrenic nerve palsy
4. Intraventricular hemorrhage (IVH) grade III or IV
5. Absence of informed consent
6. Out born infants

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure | 72 hours
  1. Treatment failure during the first 72 hours post-extubation.
  2. Reintubation (failure of extubation) within 72 hours' post extubation.
  Treatment failure is defined as:
  * Hypoxia (FiO 2 requirement > 0.35)
  * Respiratory acidosis defined as pH < 7.2 & PCo2> 60 mmHg
  * Major apnea requiring mask ventilation or > 4 episodes/ hour.
  The protocol will discontinue according to treatment failure criteria as mentioned above.
  Rescue treatment with NIPPV will be allowed and will be considered as treatment failure

SECONDARY OUTCOMES:
Death prior to discharge | 90 days from birth
  Death
Intraventricular haemorrhage IVH (grades III & IV) | 7 days after extubation
  defined as haemorrhage causing ventricular dilatation with or without brain parenchymal involvement
Pneumothorax | 7 days after extubation
  diagnosed radiologically
Bronchopulmonary dysplasia (BPD) | 36 weeks' postmenstrual age
  defined as requirement for supplemental oxygen at 28 days of life or requirement for supplemental oxygen at 36 weeks' postmenstrual age
Necrotizing enterocolitis | 7 days after extubation
  defined according to modified Bell's criteria (stage 2 to 3)
Gastrointestinal perforation | 7 days after extubation
  diagnosed radiologically or at operation
Nosocomial sepsis | 7 days after extubation
  defined as positive blood or cerebrospinal fluid (CSF) cultures taken after five days of age
Retinopathy of prematurity (ROP) | 40 weeks corrected postnatal age
  stage 3 or greater (International classification)
Duration of hospitalisation or Length of stay (in days) | From admission to first discharge from hospital, assessed up to 6 months
  Number of days in hospital until first discharge

CONTACTS AND LOCATIONS:
Overall Officials: Raniah Aljeaid, Principal Investigator — King Fahad Armed Forces Hospital Jeddah; Nisreen Kafi, Study Director — King Fahad Armed Forces Hospital Jeddah; Fawzia Sabbagh, Study Director — King Fahad Armed Forces Hospital Jeddah; Mai Abu Seoud, Study Chair — King Fahad Armed Forces Hospital Jeddah
Locations (1):
- King Fahad Armed Forces Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lee J, Kim HS, Jung YH, Shin SH, Choi CW, Kim EK, Kim BI, Choi JH. Non-invasive neurally adjusted ventilatory assist in preterm infants: a randomised phase II crossover trial. Arch Dis Child Fetal Neonatal Ed. 2015 Nov;100(6):F507-13. doi: 10.1136/archdischild-2014-308057. Epub 2015 Jul 15. PMID 26178463
- [Result] Stein H, Howard D. Neurally adjusted ventilatory assist in neonates weighing <1500 grams: a retrospective analysis. J Pediatr. 2012 May;160(5):786-9.e1. doi: 10.1016/j.jpeds.2011.10.014. Epub 2011 Dec 3. PMID 22137670

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03388437/Prot_SAP_000.pdf